CLINICAL TRIAL: NCT03636724
Title: Evaluation of an E-intervention on Multiple Health Behaviour Change for Chinese Cardiac Patients in Home-based Rehabilitation
Brief Title: Evaluation of an E-intervention on MHBC for Chinese Cardiac Patients in Home-based Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yanping DUAN, Assistant Professor, Dr. Duan, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FRG2/17-18/099
Record Dates: First submitted 2018-08-02; First posted 2018-08-17 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Cardiac Rehabilitation; Physical Activity; Fruit and Vegetable Intake
Keywords: E-health intervention; multiple health behavior change; Health Action Process Approach Model; Cardiac patients
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients will receive the interventions on both PA and FVI simultaneously.
  Interventions: Behavioral: E-intervention
- Waiting control group (No Intervention): Patients will not receive any supportive interventions on PA or FVI during the intervention period but will be provided with the same intervention at follow-up six-month after the intervention.

INTERVENTIONS:
Behavioral: E-intervention — The 10-week e-health intervention will target HAPA-based social-cognitive variables of PA and FVI. Particularly, Week 1: risk perception and outcome expectancies; Week 2: goal setting; Week 3: development of action plans; Week 4: revision and adjustment of previous action plans; Week 5: development of coping plans; Week 6: revision and adjustment of previous coping plans; Week 7: development of perceived social support; Week 8: revision and adjustment of previous social support. Week 9-10: self-monitoring. Self-efficacy will be a fixed intervention variable involved from week 2 to week 10. Additionally, some behaviour change techniques will be employed in the intervention in order to facilitate the implementation and maintenance of behaviour.
  Arms: Intervention group

SUMMARY:
By using the Health Action Process Approach (HAPA) model as a theoretical backdrop, the proposed study aims to provide a 10-week e-health learning strategies for Chinese cardiac patients, with which they can follow at home after rehabilitation discharge. The current study will examine whether the cardiac rehabilitation patients in intervention group would increase their physical activity (PA) level and fruit-vegetable intake (FVI), improve the social-cognitive variables of PA and FVI, and enhance mental health outcomes in comparison with control condition; and whether the social-cognitive variables would mediate the association between intervention and adopting a healthy lifestyle. The study findings may contribute to the current multiple health behaviour intervention research and support Chinese cardiac patients to maintain rehabilitation outcomes and cultivate a healthy lifestyle.

DETAILED DESCRIPTION:
For the main study, the sample size will be estimated by using G*Power 3.1 software with MANOVA of repeated measures approach. For achieving a medium effect size of 0.25 (Duan et al., 2017), with a power (1-β) of 0.8 and an alpha of 0.05, the total sample size will be 116. Assuming a dropout rate of approximately 30%, a total of 166 participants will be required for the study evaluation.

All data will be analyzed by using SPSS 23.0 software. Independent samples t-tests and Chi2-tests will be adopted to examine the characteristics of drop out and compare the differences of baseline data at T1. Statistical significance will be set at 5% level (two-tailed). The intervention effects on behavioural, social-cognitive and mental health status-related indicators will be tested by conducting the multivariate analysis of variance (MANOVA) with repeated measures, with time (T1, T2 and T3) as the with-in subjects factor and group (IG and CG) as the between-subjects factor. Missing data will be imputed within each measurement point in time using the Expectation-Maximization (EM) method. Furthermore, the intervention effect on healthy lifestyle indicator will be examined by performing a multinomial logistic regression model. The multiple-mediator model will be conducted to test the mediation effects with the use of SPSS macro (Preacher & Hayes, 2008).

ELIGIBILITY:
Inclusion Criteria:

* no restriction of physical mobility under the cardiac function at entry
* no restriction of relevant diseases such as diabetes or fruit allergies
* As the study involves an online website and mobile phone SMS, only participants with access to the Internet via mobile phone will be enrolled

Exclusion Criteria:

* have restrictions of physical mobility under the cardiac function at entry
* have restrictions of relevant diseases such as diabetes or fruit allergies
* cannot use the Internet and mobile phone

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2021-07-31 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change of weekly amount of physical activity (PA) | From baseline to the 9th week (at the end of intervention) and 3-month follow-up
  The level of PA will be measured through the short Chinese version of the International Physical Activity Questionnaire (IPAQ-C) questionnaire. Participants will be asked to estimate the number of days and hours spent for vigorous, moderate and walking activities during the past week. The total physical activity score for each participants is the sum of frequency per week, multiplied by time-consumption (minutes) each time.
Change of daily portions of fruit-vegetable intake (FVI) | From baseline to the 9th week (at the end of intervention) and 3-month follow-up
  Fruit and vegetable intake (FVI) will be measured with four items, including fruit or vegetable juice, fruit, cooked or steamed vegetables, and raw vegetables. Respondents will be asked to count the number of portions of fruit and vegetables they consumed on average during a typical day. Each item has 11 options for the number of portions such as 0, 0.5, 1, 1.5, 2, 2.5, ..., and 5 or above. The total portion of fruit and vegetable consumption is the sum of each item.

SECONDARY OUTCOMES:
Change of self-efficacy of PA and FVI | From baseline to the 9th week (at the end of intervention) and 3-month follow-up
  Self-efficacy will be assessed with three dimensions consisting of motivational, maintenance and recovery self-efficacies with the stem "I am certain that…" followed by 5 items for PA such as "…I can be physically active permanently at a minimum of 5 days a week for 30 minutes even if it is difficult", or followed by 5 items for FVI such as "…I can eat 5 portions of fruit and vegetable a day even if it is difficult." Answers will be given on a 5-point Likert scale, ranging from don't agree at all "1" to agree completely "5". The mean value of the total score will be calculated and the higher score denotes to the higher level of self-efficacy.
Change of intention of PA and FVI | From baseline to the 9th week (at the end of intervention) and 3-month follow-up
  The intention for PA will be assessed with the stem "I intend to do for at least 30 minutes a day on minimum 5 days a week or at least 150 minutes a week with…" followed by 3 items such as "… vigorous sport", "…moderate PA" and "…mild PA". The intention for FVI will be measured by the stem " I seriously intend to..." followed by 3 items such as "eat at least 5 servings of fruit and vegetable each day" and "… drink each day at least one glass of fruit or vegetable juice". Answers will be given on a 4-point Likert scale, ranging from not true "1" to exactly true "5". The mean value of the total score will be calculated and the higher score denotes to the higher level of intention.
Change of planning of PA and FVI | From baseline to the 9th week (at the end of intervention) and 3-month follow-up
  Planning indicator will be assessed with 6 items, consisting of action planning and coping planning with 3 items for each dimension. The item of action planning for PA will be asked such as "…which concreted PA I will pursue", for FVI such as "…how I will prepare the food". The items of coping planning for PA will be asked such as "…how I can stay active, even if something happened", for FVI such as "what I can do in difficult situations, in order to remain true to my own resolutions". Answers will be given on a 5-point Likert scale, ranging from totally disagree "1" to totally agree "5". The mean value of the total score will be calculated and the higher score denotes to the higher level of planning.
Change of perceived social support of PA and FVI | From baseline to the 9th week (at the end of intervention) and 3-month follow-up
  For the perceived social support, the scale will be measured with the stem as "How do you perceived your environment?" followed by 3 items for PA such as"….People like my friends help me to stay physically active", or followed by 3 items for FVI such as "…People like my friends help me to eat healthily". Answers will be given on a 4-point Likert scale, ranging from totally disagree "1" to totally agree "5". The mean value of the total score will be calculated and the higher score denotes to the higher level of perceived social support.
Change of perceived quality of life: WHO Quality of Life-BREF | From baseline to the 9th week (at the end of intervention) and 3-month follow-up
  This indicator will be assessed by using the short version of the World Health Organisation Quality of Life (WHOQOL-BREF). Respondents will be first asked about their general quality of life as "How would you rate your quality of life?", then 7 items in physical health sub-domain will be used, such as the example item "To what extent do you feel that physical pain prevents you from doing what you need to do?". Answers will be given on a 5-point Likert scale, ranging from very poor "1" to very good "5". The mean value of the total score will be calculated and the higher score denotes to the higher level of perceived quality of life.
Change of depression | From baseline to the 9th week (at the end of intervention) and 3-month follow-up
  Level of depression will be assessed with the use of the Center for Epidemiologic Studies Short Depression Scale (CES-D 10). Respondents will be asked with the stem as "In the past week how often I feel …" followed by 10 items such as "…I was bothered by things that usually don't bother me". Answers will be given on a 4-point Likert scale, ranging from rarely or none of the time (less than 1 day) "0" to most or all of the time (5-7 days) "3". The mean value of the total score will be calculated and the higher score denotes to the higher level of depression.
Change of body mass index (BMI) | From baseline to the 9th week (at the end of intervention) and 3-month follow-up
  Participants will be asked to report their body height (in m) and body weight (in kg) for calculating the BMI, using the equation "BMI=weight/ height square".

OTHER OUTCOMES:
Social-demographic information | At the beginning of intervention (Baseline)
  The items consist of gender, age, marital status, education level, rehabilitation treatment history, and current work status.

CONTACTS AND LOCATIONS:
Overall Officials: Yanping Duan, Principal Investigator — Hong Kong Baptist University
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duan Y, Li X, Guo L, Liang W, Shang B, Lippke S. A WeChat Mini Program-Based Intervention for Physical Activity, Fruit and Vegetable Consumption Among Chinese Cardiovascular Patients in Home-Based Rehabilitation: A Study Protocol. Front Public Health. 2022 Mar 22;10:739100. doi: 10.3389/fpubh.2022.739100. eCollection 2022. PMID 35392478

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT03636724/Prot_SAP_002.pdf
  • Informed Consent Form (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT03636724/ICF_001.pdf